CLINICAL TRIAL: NCT06886750
Title: Investigation of Waning Time in Patients with Cervical Dystonia Converted to Botulinum Toxin a
Brief Title: The Effects of Waning of Botulinum Toxin in the Treatment of Cervical Dystonia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Manjog Enterprises Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dysportstudy1
Record Dates: First submitted 2025-02-20; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Cervical Dystonia, Primary
Keywords: botulinum toxin injections; waning effect; dystonia
MeSH Terms: conditions — Cervical Dystonia, Primary; Dystonia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Single blind study
Who Masked: Participant
Masking Description: Patinet blinded to the toxin type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aboBoNT-A (Active Comparator): 1. Next 3 injections (every 12 weeks) are using aboBoNT-A (Dysport)
  2. First Dysport injection: 1:2.5 ona/incoBoNT-A: aboBoNT-A dose ratio conversion (reconstitution is 2 ml in a 500 U aboBoNT-A vial) (V1)
  3. Second and third injection: clinical optimization of aboBoNT-A dosing pattern at 12-weeks post aboBoNT-A injection. (V2 and V3). The 12 week period is compulsory.
  4. Return to original BoNT-A formulation (1:2.5 ona/incoBoNT-A: aboBoNT-A dose ratio), using same injection pattern as V3 (V4)
  5. Non-injection final study visit to conduct all assessments (V5)
  Interventions: Drug: Botulinum toxin type A injection
- Original toxin arm (Active Comparator): 1. Next 3 injections (every 12 weeks) are the same toxin as the original
  2. First injection: Dose may be optimized as per the investigators discretion or kept the same (reconstitution is 1 ml in a 100 U ona/incoBoNT-A vial) (V1)
  3. Second and third injection: clinical optimization of the dose as required with dosing pattern at weeks 12 post injection. (V2 and V3). The 12 week period is compulsory.
  4. Continue with the original toxin, using same injection pattern as V3 (V4)
  5. Non-injection final study visit to conduct all assessments (V5)
  Interventions: Drug: Botulinum toxin type A injection

INTERVENTIONS:
Drug: Botulinum toxin type A injection — Injection of toxin

SUMMARY:
The main treatment for cervical dystonia is botulinum toxin injections. However, some patients receiving this treatment after many years tend to experience short duration of benefit. Typically, botulinum toxin brands used in clinic are Botox or Xeomin. Another type of botulinum toxin is called Dysport (Ipsen Biopharmaceuticals), and Dysport may increase duration of benefit from the injections. The study is selecting patients from the investigator's clinics who are not satisfied with the duration of their treatment and are willing to switch to Dysport and the investigators will monitor if Dysport will increase the duration of benefit over a total of 3 treatments. A group of patients will be switched to Dysport while another group will remain on their original botulinum toxin formulation. The patients will be unaware of the treatment switch and hence are considered to be blinded. The investigators will not be blinded. Treatments are given every 3 months. All study visits will occur at the local sites of the 3 recruiting sites.

DETAILED DESCRIPTION:
Cervical dystonia (CD) is a disabling and often painful condition clinically characterized by abnormal neck and head postures and movements often associated with tremor and chronic pain. Botulinum toxin type A (BoNT-A) is an effective and safe ﬁrst-line therapy for CD. However, in a recent patient perspective survey, symptom re-emergence between injections (a mean 10.5 weeks) was reported in 88% of patients with a waning time of ≤8 weeks in one-third of patients. Waning treatment effects prior to re-injection reduces quality of life as 47% of patients are somewhat satisﬁed, and 39% were not satisﬁed with their therapy as symptoms may follow a "yo-yo" pattern . 45% of patients would prefer a ≤10-week treatment cycle due to the short therapeutic response. However, practicality of injecting patients more frequently and concerns about potential immunologically mediated resistance to BoNT-A has resulted in a standard of treating at intervals of at least 12 weeks. Thus, a signiﬁcant unmet need is a long-lasting therapy that delays symptom re-emergence and may improve patient satisfaction and outcomes.

Nine published clinical studies have studied the direct comparison between Botox and Dysport in CD patients and authors concluded that a simple dose-conversion factor is not applicable as the ratio for Botox to Dysport was extremely variable, ranging from 1.2 to 13.3. Yun et al demonstrated that conversion to Dysport using a Botox:Dysport ratio of 1:2.5 was not inferior to Botox. A double blind, crossover study lasting 3 injection cycles studied 2 ratios (1:3 and 1:4) and found at both conversion ratios, Dysport was superior to Botox in terms of symptom reduction and duration of effect, although higher frequency of adverse effects such as dysphagia was reported. More recently, a double-blind, randomized crossover study evaluated 2 conversion ratios (1:3 and 1:1.7) that did not show any differences in efficacy in the short term, but the effect of Botox was reduced after 3 months. At week 12, a statistically significant difference in efficacy between abobotulinumtoxinA and onabotulinumtoxinA (1:3) was observed, suggesting a shorter duration of effect for the latter when this ratio (at low dose) was used. Thus, in this research study, the objective is to determine if conversion ratio of 1:2.5 (Botox:Dysport) from the patient's optimized, stable treatment (either Botox or Xeomin) can increase duration of BoNT-A efficacy.

A pilot study published by our research group reported a significant increase in waning time and efficacy following the conversion to aboBoNT-A in 27 CD patients who had a waning time of ≤8-weeks on their original BoNT-A formulation (either onaBoNT-A/incoBoNT-A). The results of the pilot study were limited by the lack of participant blinding and absence of a control group. Thus, a randomized, controlled, single-blind study will be conducted to determine whether the conversion to aboBoNT-A affects waning time, clinical outcomes and treatment satisfaction in patients experiencing early waning with ona/incoBoNT-A.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above with a diagnosis of isolated CD
* Experience efficacious relief with a waning time of ≤8 weeks post-injection
* Must have received the same dose and injection pattern of onaBoNT-A or incoBoNT-A for at least 3 injection cycles prior to study initiation with an injection cycle of 12 weeks

Exclusion Criteria:

* Require a total dose <80 U or >300 U ona/incoBoNT-A
* Pure reterocollis or suspected secondary non-responsiveness
* No interest in switching between BoNT-A formulations
* Prolonged history of dysphagia
* History of poor response to BoNT-A or BoNT-B
* Inability to complete study visits or sign informed consent
* Pregnancy
* Known resistance or contradictions to any BoNT-A
* Known hypersensitivity to BoNT-A or related compound

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Waining time. | At the end of each cycle for 3 cycles. Each cycle is 12 weeks in duration as the reinjection is done every 12 weeks.
  Waning time - time from last injection to participant perception of treatment effects starting to wear off. An increase in waning time is a better outcome. Values will be between 8 to 12 weeks.

SECONDARY OUTCOMES:
• Modified Tsui Scale | At the end of each cycle for 3 cycles. Each cycle is 12 weeks in duration as the reinjection is done every 12 weeks.
  • Modified Tsui Scale for assessment of severity of cervical dystonia. A lower score is an improvement in outcome. Minimum value is 0 and maximum value is 18.
• 5-point Likert participant reported treatment satisfaction tool | At the end of each cycle for 3 cycles. Each cycle is 12 weeks in duration as the reinjection is done every 12 weeks.
  • 5-point Likert participant reported treatment satisfaction tool of injection of botulinum toxin for cervical dystonia. . A higher score on the scale denotes an improvement in the symptoms of cervical dystonia. Minimum value is 0 and maximum value is 5.
• Onset of treatment relief using the symptom tracker | At the end of each cycle for 3 cycles. Each cycle is 12 weeks in duration as the reinjection is done every 12 weeks.
  • Onset of treatment relief using the symptom tracker. This is the time at which point improvement in the symptoms of cervical dystonia are noted by the participant.
• Safety of the use of botulinum toxin injection for cervical dystonia | At the end of each cycle for 3 cycles. Each cycle is 12 weeks in duration as the reinjection is done every 12 weeks.
  • Safety will be measured as reported side effects by the patient from the injection of botulinum toxin for cervical dystonia. Treatment related adverse events will be documented and commented upon as related or unrelated to the treatment. This will be documented at every 12 week clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — Univ of Western Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samotus O, Jog M. Conversion to AbobotulinumtoxinA Increases Waning Time and Efficacy for Cervical Dystonia. Mov Disord Clin Pract. 2023 Mar 1;10(5):756-763. doi: 10.1002/mdc3.13696. eCollection 2023 May. PMID 37205243